CLINICAL TRIAL: NCT05254639
Title: Evaluation of the Efficacy of Donepezil in the Treatment of Oxaliplatin-induced Peripheral Neuropathy: Proof of Concept Study
Brief Title: Donepezil for Oxaliplatin-induced Neuropathy Peripheral Neuropathy: Proof of Concept Study
Acronym: DONEPEZOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC K 2020 PEZET; 2021-005326-23 (EudraCT Number)
Record Dates: First submitted 2022-02-04; First posted 2022-02-24 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Digestive Oncology; Supportive Care
Keywords: Pharmacology; Chronic Pain; Oxaliplatin; Chemotherapy-induced peripheral neuropathy; Donepezil
MeSH Terms: conditions — Chronic Pain | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donepezil (Experimental): 5 mg/day for 4 weeks then 10 mg/day for 12 weeks
  Interventions: Drug: DONEPEZIL
- Placebo (Placebo Comparator): 5 mg/day for 4 weeks then 10 mg/day for 12 weeks
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: DONEPEZIL — 5 mg daily for 4 weeks + 10 mg daily for 12 weeks according to tolerance or efficacy
  Arms: Donepezil
Drug: PLACEBO — 5 mg daily for 4 weeks + 10 mg daily for 12 weeks according to tolerance or efficacy
  Arms: Placebo

SUMMARY:
The use of oxaliplatin in the treatment of colorectal or pancreas cancer induces (>75% of patients) severe sensorimotor neuropathy decreasing the quality of life of cancer survivors. Today, no treatment remains univocal for these peripheral neuropathies. But preclinical works have demonstrated that donepezil (acetylcholinesterase inhibitor use for Alzheimer's disease) was able to prevent and treat neuropathic symptoms in oxaliplatin-treated rats.

Present study aims to assess the therapeutic efficacy of donepezil on oxaliplatin-induced peripheral neuropathy (OIPN) in cancer survivors. Bibliographic data suggests an antineuropathic effect of donepezil in human and animal models. In clinic, a study have shown in healthy volunteers that donepezil (associated with gabapentin) reduced the pain threshold (better than gabapentin alone) caused by stimulation of the sural nerve, without severe adverse effect. Similarly, two studies in patients with neuropathic pain demonstrated that donepezil increases analgesic effect of gabapentin. Finally, a case report demonstrated an analgesic effect of donepezil in painful Alzheimer's disease patients. In animals, several studies demonstrated that donepezil induces analgesic and neuroprotective effects. Recently, a preclinical study demonstrated that donepezil induced antineuropathic effect in diabetic mice with neuropathic pain. Research unit INSERM U1107 (partner of the DONEPEZOX study) demonstrated the antineuropathic effects of donepezil in several animal models of chemotherapy-induced peripheral neuropathies, and very recently, a study have confirmed these results with oxaliplatin and cisplatin. These clinical and preclinical data have thus highlighted the potential beneficial effect of donepezil on neuropathic symptoms, without any significant adverse effects. Therefore the hypothesis is that the use of donepezil could reduce the symptoms of OIPN, limit the decrease in quality of life and the appearance of comorbidities (anxiety/depression) in cancer survivors.

For this purpose, the investigators propose here a proof of concept, multicentre, phase II, randomised, double-blind, placebo-controlled clinical study. The primary objective will be the curative efficacy of donepezil on the severity of OIPN in patients who have completed oxaliplatin-based chemotherapy for the treatment of colorectal or pancreas cancer and have peripheral neuropathy of grade ≥2. This will be assessed using the EORTC QLQ-CIPN20 sensory scale. Our methodological choice to use the QLQ-CIPN20 as the primary endpoint will allow us to more accurately (and in a standardized manner) characterize neuropathic symptoms and assess the therapeutic effect of donepezil on these symptoms. In addition, as secondary objectives, we will study the effect of donepezil on neuropathic pain, the intensity of neuropathic symptoms, health-related quality of life, and the tolerance of donepezil.

The 80 patients required will be randomized (1:1) to receive either placebo or donepezil (5 mg daily for 4 weeks and then 10 mg daily for 12 weeks as a single dose and according to tolerance and efficacy). Patients will be followed for 1 month after the end of treatment to assess the OIPN. As a proof of concept study, responder rate will be assessed only for Donepezil arm (primary objective) and compared between each treatment arm (secondary objective) after a minimum of 12 weeks of treatment. A responder will be defined as a patient with a decrease of neuropathic grade according to CIPN20 sensory score compraed to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received chemotherapy with oxaliplatin for all stage of colorectal or pancreas cancer,
* QLQ-CIPN20 sensory score ≥30,
* Diagnosis of chemotherapy-induced peripheral neuropathy treated or not by stable antineuropathic/analgesic treatment (opioids, pregabalin, gabapentin, duloxetine and other antidepressants or anticonvulsants) for at least 1 month,
* Chemotherapy completed for at least 6 months,
* Patients affiliated to the French national health insurance,
* Written informed consent,
* French language comprehension.

Exclusion Criteria:

* Cancer relapse or secondary cancer,
* Lack of effective contraception in patients (female) of childbearing age, pregnant or breastfeeding women, women of childbearing age who have not taken a pregnancy test,
* Patient with a chronic progressive disease with associated chronic pain (excluding oxaliplatin-induced peripheral neuropathy),
* Diabetic patient (excluding non-insulin- or insulin-treated diabetes less than 5 years old) or presence of proven diabetic neuropathy,
* Other types of neuropathies,
* ALT / AST elevated more than 3 times the normal values,
* Severe cardiovascular disease (as determined by clinician), bradycardia (< 55 bpm), cardiac conduction disorders such as sinus disease or other supraventricular conduction abnormalities such as sino-auricular or atrioventricular block (assessed by electrocardiogram),
* History of peptic ulcer disease or active peptic ulcer disease,
* Asthma or chronic obstructive pulmonary disease,
* Known allergy to donepezil or piperidine derivatives,
* Known galactose intolerance, known Lapp lactase deficiency or known glucose or galactose malabsorption syndrome (rare hereditary diseases),
* Drug interactions: CYP3A4 inhibitors (ketoconazole, itraconazole and erythromycin); CYP2D6 inhibitors (fluoxetine, quinidine) and enzymatic inducers (rifampicin, phenytoin, carbamazepine),
* Known dependence on alcohol and/or drugs,
* Known psychotic disorders, patient under antipsychotics,
* Planned surgery during the trial,
* Impossible to undergo the medical follow-up of the trial for geographical, social or psychological reasons,
* Person under guardianship, curatorship, safeguard of justice or person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire-Chemotherapy Induced Peripheral Neuropathy 20 (QLQ-CIPN20) | through study completion, an average of 4 months.
  A self-reported questionnaire, consisting of 20 questions which assess the symptoms and functional limitations of CIPN from the patients' perspective. The questionnaire is divided in 3 subscales: sensory, motor, and autonomic and gives a comprehensive picture of the nature, frequency, and severity of CIPN.
  For each subscale and for the entire questionnaire, a score from 0 to 100 is generated. The higher the score, the more severe the neuropathic symptoms.

SECONDARY OUTCOMES:
11-point pain Numeric Rating Scale (NRS) | through study completion, an average of 4 months
  The NRS is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. The score of 0 = No pain and 10 = worst possible pain.
Douleur Neuropathique-4 (DN4) interview | At inclusion
  The interview portion of the DN4 questionnaire is a clinician-administered screening tool for neuropathic pain.
  The questionnaire includes 7 items, grouped into two questions. Each item, is answered as either YES or NO.
  A final cumulative patient's score is obtained by allocating 1 point for each YES and 0 point for each NO. If the patient's score ≥3/7, the test is positive.
  This evaluation will be carried out only if the 11-point pain NRS ≥4/10.
Neuropathic Pain Symptoms Inventory (NPSI) | through study completion, an average of 4 months.
  This self-reported questionnaire assesses different neuropathic pain symptoms. The French NPSI includes 12 items that discriminates and quantifies five distinct dimensions of neuropathic pain.
  This evaluation will be carried out only if the 11-point pain NRS ≥4/10.
Quality of Life Questionnaire-Cancer 30 (QLQ-C30) | through study completion, an average of 4 months.
  This EORTC self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
Hospital Anxiety and Depression scale (HADS) | through study completion, an average of 4 months.
  This self-reported questionnaire permits to detect anxiety and depressive disorders. There are 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and 7 to the depressive dimension (total D), thus obtaining two scores (maximum score of each score = 21). To detect anxiety and depressive symptoms, the following interpretation is proposed for each of the scores (A and D):
  * ≤7: absence of symptomatology
  * 8 to 10: suspicious symptomatology
  * ≥11: certain symptomatology
Patients' Global Impression of Change (PGIC) | 4 months
  PGIC is aimed at assessing the general effectiveness of the treatment. This scale consists of 7 level descriptors answering the question "How are you?" distributed in three ways: (i) improved (very/medium/slightly), (ii) unchanged and (iii) aggravated (slight/medium/very).

CONTACTS AND LOCATIONS:
Overall Officials: Denis PEZET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (34):
- France (34):
  - Hôpital privé d'Antony, Antony
  - CH d'Argenteuil, Argenteuil
  - CHU de Besançon, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier du Cotentin, Cherbourg
  - Centre Hospitalier Public du Cotentin, Cherbourg
  - CH de Cholet, Cholet
  - CHU clermont-ferrand, Clermont-Ferrand
  - Centre Hospitalier Compiègne-Noyon, Compiègne
  - Clinique de Flandre, Coudekerque-Branche
  - CHU de Dijon Bourgogne, Dijon
  - Institut de Cancérologie de Bourgogne - GRReCC, Dijon
  - CHD de Vendée, La Roche-sur-Yon
  - CH Le puy, Le Puy-en-Velay
  - Hôpital Franco-Britanique, Levallois-Perret
  - chu de Limoges, Limoges
  - CH Saint Joseph Saint Luc, Lyon
  - Clinique de la sauvegarde, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Hopital Saint Joseph de Marseille, Marseille
  - Hôpital Européen de Marseille, Marseille
  - Groupe Hospitalier des Portes de Provence, Montélimar
  - Hôpital Saint-Louis - AP-HP, Paris
  - Hôpital Privé des Cotes d'Armor, Plérin
  - CHU de Poitiers, Poitiers
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - CHU de Reims, Reims
  - Institut Godinot, Reims
  - CHU de Saint-Etienne, Saint-Etienne
  - Institut de Cancérologie Paris Nord, Sarcelles
  - Groupe Hospitalier Saint Vincent - Clinique Saint Anne, Strasbourg
  - CHU de Bordeaux, Talence
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon
  - CH de Valence, Valence

REFERENCES:
- [Derived] Kerckhove N, Tougeron D, Lepage C, Pezet D, Le Malicot K, Pelkowski M, Pereira B, Balayssac D. Efficacy of donepezil for the treatment of oxaliplatin-induced peripheral neuropathy: DONEPEZOX, a protocol of a proof of concept, randomised, triple-blinded and multicentre trial. BMC Cancer. 2022 Jul 7;22(1):742. doi: 10.1186/s12885-022-09806-8. PMID 35799138